CLINICAL TRIAL: NCT03442998
Title: Walking Green: Developing an Evidence-base for Nature Prescriptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1703S09101
Record Dates: First submitted 2017-07-19; First posted 2018-02-22 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Stress; Attention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suburban (Other): Study participants will wall on a suburban sidewalk setting for 50 minutes.
  Interventions: Other: Suburban walk
- Nature (Other): Study participants will wall on a nature path setting for 50 minutes.
  Interventions: Other: Nature walk

INTERVENTIONS:
Other: Suburban walk — Each subject is tested under the 'suburban' condition. We will compare the stress response and working memory response to walking in the two experimental conditions ((1)response to walking on a nature path and (2) response to walking on an urban sidewalk).
  Arms: Suburban
Other: Nature walk — Each subject is tested under the 'nature' condition. We will compare the stress response and working memory response to walking in the two experimental conditions ((1)response to walking on a nature path and (2) response to walking on an urban sidewalk).
  Arms: Nature

SUMMARY:
The investigators hypothesize that walking on a nature trail will lead to greater reductions in stress and greater improvements in the capacity to direct attention as compared to walking on a suburban sidewalk.

The effects of walking in these different locations will be measured using physiological and psychological outcomes. The study design is a randomized with-in person cross-over trial. Subjects will take six 50-minute walks, one walk per week for six weeks. Three walks will occur in the urban setting and three in the nature setting. The order of the conditions will be randomly assigned to each subject, so that half of the subjects will complete the urban walks first and half the subjects will complete the nature walks first. There will be a two-week washout period between the two sets of walks. Day of the week will be fixed within person, and walks will occur during the mild weather months. In the case of inclement weather, the weekly walk will be skipped and an additional week will be added to the schedule. Limiting the frequency to one walk per week maximizes feasibility of the protocol and minimizes training effects, with any training effects over time being handled primarily by randomization (condition order is balanced), but also in the statistical analysis.

DETAILED DESCRIPTION:
Suburban walks will be mapped out in clean, safe streets with sidewalks within 3 miles of the Arboretum, in Chaska, Minnesota. A loop covering approximately 1.25 miles will be mapped. At a usual walking speed of 20 minutes per mile, a subject will complete ~ 2 loops. Each walk will be timed so that walking speed can be included in the statistical analysis as an important covariate.

Nature Walks will take place at the University of Minnesota Landscape Arboretum, which is part of the College of Food, Agricultural and Natural Resource Sciences at the University of Minnesota. The Arboretum features more than 1,215 acres of natural landscapes with over 12 miles of trails. Subjects in this study will take their nature walks on the Green Heron Pond Trail and adjacent trails that can be connected to create a walking loop of ~1.25 miles, or an out-and-back course, matching the distance of the suburban walk. Heron Pond and its adjacent marsh and bog represent three naturally occurring ecosystems in Minnesota that are part of the state's geologic and landscape heritage. The bog trail passes through the most diverse ecotypes of any Arboretum hike. Oak woods, maple woods and the mosaic of intermingled wetlands along the boardwalk offer rich rewards for birders, school groups and families.

The primary approach to the statistical analysis will be a repeated measures multivariable linear regression model. The outcomes will be the psychological and physiological measures of stress. The primary independent variable of interest is condition (suburban v. nature). The interaction of condition and time (week of the study) provides a formal test of intervention effects (differences between the urban and nature walks). That is, over the time course of the interventions, are there significant differences in the outcomes between the urban and nature walks? Covariates to be evaluated in the models as possible confounders include the order of the conditions (urban first v. nature first), age, gender, body mass index, and overall habitual physical activity. On an exploratory basis, the investigators will test whether these covariates also serve as modifiers of the intervention effect.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 59
* No contraindications to physical activity
* No major chronic diseases or specific medications that would contraindicate exercise or potentially blunt heart rate variation during exercise

Exclusion Criteria:

* Cardiovascular disease medication
* Arthritis
* Steroids
* Certain blood pressure medications
* Diabetes
* Cancer
* Self-reported depression or anxiety / taking medication for depression or anxiety,
* Outside age range
* Inability to follow schedule including travel to arboretum
* Exceeding physical activity recommendations (250 minutes per week)
* Contraindications to walking

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability | Measurements will be made at baseline one-week before the first walk, immediately before and after each walk, and within three days following the third walk of each condition (nature vs suburban).
  High frequency heart rate variation using ambulatory heart rate monitors (milliseconds).
Change in Blood Pressure | Measurements will be made at baseline, immediately before and after each walk of each condition (nature vs suburban).
  Blood pressure (mmHg) using a standard blood pressure cuff.
Change in Cortisol Dynamics | Measurements will be made before each walk of each condition (nature vs suburban).
  Diurnal cortisol dynamics measured by salivary cortisol (ug/dl), as the normal drop in cortisol during the day is attenuated by exposure to chronic stress.
Change in Cytokine Blood Concentration | Measurements will be made before each walk of each condition (nature vs suburban).
  Pro- and anti-inflammatory cytokine concentrations in blood (pg/mL), as stress typically induces an inflammatory response. Blood samples are collected by pricking the subject's finger-tip, collecting drops of blood on Protein SaverTMpaper (Whatman) and then drying the blood spots. The dried blood spots (DBS) are frozen and stored until assayed.
Change in Attention restoration | Measurements will be made at baseline one-week before the first walk, immediately before and after each walk, and within three days following the third walk of each condition (nature vs suburban).
  The Backward Digit Span test is one of the oldest tests used to evaluate working memory and is used to assess capacity to direct attention (i.e., attention restoration).
Change in CESD | Measurements will be made at baseline, immediately before and after each walk of each condition (nature vs suburban).
  CESD: Stress is strongly associated with depression. To measure depressive symptoms we will use the Center for Epidemiological Studies Depression Scale (CESD). Scores are determined by summing the participants' answers to all 20 items from 1 ("less than 1 day") to 4 ("5-7 days") pre- and post-walk in each intervention location (nature vs suburban).
Change in PANAS | Measurements will be made at baseline, immediately before and after each walk of each condition (nature vs suburban).
  PANAS: Stress is associated with decreased positive and increased negative affect (mood). We will measure affect using the Positive and Negative Affect Scale (PANAS).
  Scores are determined by summing the participants' answers to all 20 items from 1 ("very slightly or not at all") to 5 ("extremely") pre- and post-walk in each intervention location (nature vs suburban).
Change in STAI | Measurements will be made at baseline, immediately before and after each walk of each condition (nature vs suburban).
  Anxiety: Stress is associated with increased levels of anxiety. Anxiety will be measured using the State and Trait Anxiety Inventories (STAI). Scores are determined by summing the participants' answers to all 20 items from 1 ("not at all") to 4 ("frequently so") pre- and post-walk in each intervention location (nature vs suburban).
Change in Perceived stress | Measurements will be made at baseline, immediately before and after each walk of each condition (nature vs suburban).
  Perceived stress: Cohen's perceived stress scale (PSS) will be used to measure the extent to which subjects assess the events and situations in their lives to be stressful. Scores are determined by summing the participants' answers to all 10 items from 1 ("never") to 4 ("very often") pre- and post-walk in each intervention location (nature vs suburban).

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Pereira, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Minnesota Landscape Arboretum, Chaska, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No